CLINICAL TRIAL: NCT03022903
Title: Blue Light Photodynamic Therapy Treatment for Distal and Lateral Subungual Toenail Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Boni Elewski, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150128007
Record Dates: First submitted 2015-10-16; First posted 2017-01-18 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Toenail Onychomycosis; Distal and Lateral Subungual Toenail Onychomycosis
MeSH Terms: interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photodynamic Therapy (PDT) (Other): PDT with ALA (photosensitizer) for 3 hours
  Interventions: Procedure: Aminolevulinic Acid (ALA)

INTERVENTIONS:
Procedure: Aminolevulinic Acid (ALA) — Photosensitizing
  Other Names: ALA is a topical drug used in the administration of PDT.

SUMMARY:
This research study will evaluate the safety and efficacy of using blue light photodynamic therapy (PDT) for treating toenail fungal infections.

DETAILED DESCRIPTION:
This research study will evaluate the safety and efficacy of using blue light photodynamic therapy (PDT) for treating toenail fungal infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 19 and younger than 70 years
* Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
* Diagnosed with distal lateral subungual onychomycosis (DLSO) of the great toe with both positive potassium hydroxide (KOH) and positive culture growth of Trichophyton rubrum
* No topical treatment for DLSO in the preceding 2 weeks and no oral treatment for DLSO (itraconazole or terbinafine) in the preceding 8 weeks
* At lease 20% of target great toe nail affected

Exclusion Criteria:

* Unable to comply with the protocol (as defined y the investigator; i.e. drug or alcohol abuse or history of noncompliance)
* Patients with active nail disease that would confound evaluation of DLSO, such as psoriasis
* Patients with greater than 6 toenails affected
* Over 90% of target great toe affected
* Evidence of fingernail fungal infection
* Patients with recurrent serious infections or have been hospitalized in the preceding 6 months for infection
* Patients with known history of HIV or hepatitis B or C infection
* Patients with severe, progressive, or uncontrolled with renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurologic disease
* Any subject who, in the opinion of the investigator, will be uncooperative or unable to comply with study procedures

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects diagnosed with presence of subungual culture after 3rd treatment session | 3 weeks after baseline
  Based on presence of fungal infection from culture assessment
Number of subjects with clinical cure based on photographs after the 3rd treatment session | 3 weeks after baseline
  Based on visual assessment of photographs: presence or absence of fungal infection

SECONDARY OUTCOMES:
Compare rates of mycological and clinical cure after three treatments between two groups with different ALA incubation times | 3 weeks after baseline
Evaluate the durability of treatment outcomes with subungual culture and photographs at 24 weeks | 24 weeks after first treatment
Evaluate tolerability to treatment using a Visual Analog Scale (VAS) pain scale questionnaire at each treatment visit | 1 week after baseline
Evaluate tolerability to treatment using a Visual Analog Scale (VAS) pain scale questionnaire at each treatment visit | 2 weeks after baseline
Evaluate tolerability to treatment using a Visual Analog Scale (VAS) pain scale questionnaire at each treatment visit | 3 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Dermatology at the Whitaker Clinic, Birmingham, Alabama, United States